CLINICAL TRIAL: NCT00282841
Title: Visualization of the Cerebral Arterial Circulation Using Contrast-Enhanced Transcranial Ultrasound in Code Stroke Patients
Brief Title: Visualization of Cerebral Arteries Using Contrast-Enhanced Transcranial Ultrasound in Stroke Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated due to slow recruitment and funding ended.
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P50NS44148MATTREY; P50NS044148-06 (NIH)
Record Dates: First submitted 2006-01-26; First posted 2006-01-27 (Estimated); Results first posted 2019-08-07 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-07

CONDITIONS: Stroke
Keywords: stroke; ultrasound; occlusion; blockage; contrast solution
MeSH Terms: conditions — Stroke; Bites and Stings | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All stroke code patients (Experimental): After written informed consent Code Stroke patients will undergo a contrast-enhanced transcranial ultrasound study to visualize the intracranial arteries. To do so, an ultrasound contrast agent (Definity) will be administered intravenously and transcranial ultrasound will be applied via the temporal bone window on both sides. Goal is to visualize and assess the intracranial arteries bilaterally. This includes the following vessel segments on both sides: middle cerebral artery (M1,M2,M3 segments), anterior cerebral artery (A1,A2 segments), posterior cerebral artery (P1,P2 segments), internal carotid artery (C1/2,C3/4 segments).
  Interventions: Other: ultrasound

INTERVENTIONS:
Other: ultrasound — single intravenous administration of maximum 1.5 milliliter ultrasound contrast agent (Definity), followed by maximum 15 minutes transcranial insonation using diagnostic ultrasound.
  Other Names: Doppler

SUMMARY:
The purpose of this study is to find out more about the usefulness of ultrasound in combination with a contrast solution to look for blood vessel blockage or occlusion in the brains of stroke patients.

DETAILED DESCRIPTION:
Ischemic stroke is a common, devastating and costly disease. A stroke is usually caused by a blockage in one of the arteries that carries blood to the brain.

The purpose of this study is to visualize the blood vessels in the brain and to look for vessel occlusion (i.e., blockage) which may be the cause of stroke. Ultrasound contrast imaging may or may not improve the ability to diagnose vessel occlusion in the brain quickly and precisely, thereby expediting the therapy currently in place for acute stroke.

The contrast solutions used in this study have been approved by the Food and Drug Administration because they improve ultrasound pictures taken in the heart. While the solutions are approved for use with ultrasound in viewing the heart, the usefulness in viewing brain vessels has not been approved and is experimental.

The study will enroll 400 participants with possible diagnosis of acute stroke. Individuals participating in the study will be injected with a contrast solution via an intravenous line. A small probe will be used to obtain images of blood vessels in the head. The study researchers will measure vital signs prior to injection of the contrast solution, 5 minutes after the injection, and at the end of the ultrasound. Each participant will have a 5-minute mental function assessment and a brief neurological exam. Participants will undergo at least 3 ultrasounds. The total time of each ultrasound is less than 30 minutes.

This study is part of the Specialized Program of Translational Research in Acute Stroke to enhance and initiate translational research that ultimately will benefit stroke patients. Results from this study may help investigators learn about the future development of new diagnostic tests for stroke.

ELIGIBILITY:
Inclusion Criteria:

* patient 18 years of age or older
* code stroke patient

Exclusion Criteria:

* women with positive pregnancy test
* women who are breast feeding
* severe emphysema
* pulmonary vasculitis
* history of pulmonary emboli
* chronic renal failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2005-03; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Mattrey, MD, Principal Investigator — UCSD Stroke Center
Locations (2):
- United States (2):
  - University of California San Diego Hillcrest Medical Center, San Diego, California
  - Sharp Memorial Hospital, 7901 Frost Street, San Diego, California

REFERENCES:
- [Background] Holscher T, Sattin JA, Raman R, Wilkening W, Fanale CV, Olson SE, Mattrey RF, Lyden PD. Real-time cerebral angiography: sensitivity of a new contrast-specific ultrasound technique. AJNR Am J Neuroradiol. 2007 Apr;28(4):635-9. PMID 17416812

RESULTS

PARTICIPANT FLOW:
Groups:
- All Stroke Code Patients: Patients admitted with acute stroke code whether or not they will undergo thrombolytic therapy who received magnetic resonance angiography (MRA) or computerized tomographic angiography (CTA).
Period: Overall Study
Arm/Group | All Stroke Code Patients
Started | 61 (Anticipated recruitment 400; stopped due to funding and poor recruitment.)
Completed | 61
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Stroke Code Patients
Number analyzed (Participants) | 61
Age, Continuous [Mean (Full Range); unit: years] | 64.82 [34 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 34
Region of Enrollment [Number; unit: participants]
  United States | 61

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Visualization of the Intracranial Arteries in Comparison to Reference Method (MRA/CTA)
Description: The number of participants with successful visualization (yes/no) of the cerebral artery segments was assessed by an experienced sonographer who was blinded to the cerebral MRA/CTA.
Time Frame: within 24 hours after reference method
Population: Based on the assumption that all target intracranial vessel segments could be visualized with either one of the reference methods, CTA or MRA, in all patients enrolled, the transcranial ultrasound data was analyzed to assess how many of the target vessel segments could be visualized in comparison to the reference method.
Measure: Number; unit: participants
Units Other Than Participants: number of vessel segments visualized
Groups:
- Stroke Code Patients - Reference Method: Patients admitted with acute stroke code whether or not they will undergo thrombolytic therapy who received magnetic resonance angiography (MRA) or computerized tomographic angiography (CTA).
- Stroke Code Patients - Transcranial Ultrasound: All acute stroke patients who received magnetic resonance angiography (MRA) or computerized tomographic angiography (CTA) did receive a contrast-enhanced transcranial ultrasound study as well.
Arm/Group | Stroke Code Patients - Reference Method | Stroke Code Patients - Transcranial Ultrasound
Number analyzed (Participants) | 61 | 61
Number analyzed (number of vessel segments visualized) | 488 | 488
participants | 8 | 8

ADVERSE EVENTS:
Groups:
- Stroke Code Patients: Patients admitted with acute stroke code whether or not they will undergo thrombolytic therapy who received magnetic resonance angiography (MRA) or computerized tomographic angiography (CTA).
Arm/Group | Stroke Code Patients
Serious Adverse Events (participants affected / at risk) | 0/61
Other Adverse Events (participants affected / at risk) | 0/61

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes